CLINICAL TRIAL: NCT00006200
Title: Thalidomide and Dacarbazine for Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00096-1000; M01RR000096 (NIH)
Record Dates: First submitted 2000-09-09; First posted 2000-09-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Thalidomide; Dacarbazine

INTERVENTIONS:
Drug: thalidomide
Drug: dacarbazine

SUMMARY:
The purpose of this clinical trial is to assess the activity of thalidomide in combination with dacarbazine (DTIC) in patients with metastatic melanoma. Safety and toxicity of the two drugs will also be assessed. Dacarbazine is the standard medical treatment for metastatic melanoma. It has been shown to produce tumor shrinkage in approximately 20% of patients with advanced melanoma. This shrinkage is usually incomplete and lasts a short time. Thalidomide is a drug that inhibits tumor blood vessel growth. It can be given orally. It is hoped that this combination can be given to patients with metastatic melanoma without causing too much toxicity while increasing the response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic melanoma.
* Lesions must be measurable.
* Patient must have the following minimum labs: ANC> 1500/mm3, Hemoglobin > 8 mg/dl; platelets > 100,000 mm3; and liver function tests < 5x normal; and creatinine < 1.5 mg/dl.
* ECOG performance status > 2.
* No prior therapy with DTIC or thalidomide
* No other history of malignancy other than curatively resected basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patients must not be pregnant or lactating.
* Sexually active men and women of childbearing age must use adequate contraception. All patients must understand the potential for severe birth defects with thalidomide and must be able to follow instructions to avoid conception while taking thalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Comprehensive Cancer Center, New York, New York, United States